CLINICAL TRIAL: NCT00673270
Title: Hemodynamic and Biological Effects of Fludrocortisone and Hydrocortisone, in Healthy Volunteers With Aldosterone Induced Suppression
Brief Title: Effects of Fludrocortisone and Hydrocortisone in Healthy Volunteers With Aldosterone Induced Suppression
Acronym: AFLUCO2
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EudraCT 2007-0077969-20; CIC0203/029
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Renin Angiotensin
MeSH Terms: interventions — Fludrocortisone; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Fludrocortisone and Hydrocortisone
  Interventions: Drug: Fludrocortisone; Drug: Hydrocortisone
- 2 (Experimental): Fludrocortisone and placebo of Hydrocortisone
  Interventions: Drug: Fludrocortisone; Drug: Placebo of Hydrocortisone
- 3 (Experimental): Placebo of Fludrocortisone and Hydrocortisone
  Interventions: Drug: Hydrocortisone; Drug: Placebo of Fludrocortisone
- 4 (Placebo Comparator): Placebo of Fludrocortisone and placebo of Hydrocortisone
  Interventions: Drug: Placebo of Fludrocortisone; Drug: Placebo of Hydrocortisone

INTERVENTIONS:
Drug: Fludrocortisone — 50 µg of fludrocortisone per os
  Arms: 1; 2
Drug: Hydrocortisone — 50 mg of intravenous hydrocortisone
  Arms: 1; 3
Drug: Placebo of Fludrocortisone — Tablet of placebo of Fludrocortisone
  Arms: 3; 4
Drug: Placebo of Hydrocortisone — 2 ml of isotonic saline solution
  Arms: 2; 4

SUMMARY:
Septic shock (associated with relative adrenal insufficiency) is characterized by decreased arterial responsiveness to catecholamines. The association of hydrocortisone and fludrocortisone has demonstrated an improvement in survival in septic shock patients. If hydrocortisone has shown to increase vascular responsiveness, the role of fludrocortisone remains to be elucidated. The purpose of our study is to investigate the effect of a physiological dose of fludrocortisone and/or hydrocortisone on phenylephrine-mean arterial pressure dose-response relationship in healthy volunteers with aldosterone suppression induced by intravenous sodium loading.

ELIGIBILITY:
Inclusion Criteria:

* Men between 20 and 30 years
* Body Mass Index between 18 kg/m² and 25 kg/m²
* Normal clinical examination
* Normal biological variables
* Normal electrocardiogram and echocardiography
* Written, voluntary informed consent
* Non smoker since at least a year

Non-inclusion Criteria:

* Any history of significant allergy
* Subjects with abnormal renal, pulmonary, cardiovascular, endocrine or hepatic function
* Medication during the study
* Alcohol consumption more than 30g/day or drug addiction
* Positive serology for hepatitis B virus (HBV), hepatitis C virus (HCV) or HIV.
* Exclusion period mentioned on the Healthy Volunteers National list
* Persons deprived of freedom or under guardianship

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Phenylephrine-mean arterial pressure dose-response relationship | Between 1.5 and 3 hours after treatment

SECONDARY OUTCOMES:
Systolic and diastolic arterial pressures, heart rate, cardiac output, systemic vascular resistances | Between administration time and 24 hours after treatment
Central aortic pressures, Augmentation Index (Aix) | Between administration time and 12 hours after treatment
Arterial stiffness: Carotid-femoral Pulse Wave Velocity | Between administration time and 12 hours after treatment
Humeral diameter and distensibility | Between administration time and 12 hours after treatment
Plasma electrolytes, blood glucose, serum creatinine | Between administration time and 24 hours after treatment
Plasma renin, aldosterone, norepinephrine, epinephrine, hydrocortisone, fludrocortisone concentrations | Between administration time and 24 hours after treatment
Urinary electrolytes excretion | Between administration time and 24 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bruno LAVIOLLE, MD, Principal Investigator — Rennes University Hospital; Eric BELLISSANT, MD, PhD, Study Chair — Rennes University Hospital
Locations (1):
- Unité d'Investigation Clinique - Hôpital de Pontchaillou, Rennes, France